CLINICAL TRIAL: NCT02658773
Title: Effect of Cervical Lidocaine-prilocaine Cream on IUD Insertion Pain: A Randomized Controlled Trial
Brief Title: Lidocaine-prilocaine Cream on IUD Insertion Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LPIUD
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: IUD Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- lidocaine-Prilocaine cream (Active Comparator): lidocaine-Prilocaine anesthetic cream placed into their cervix prior to having the IUD inserted
  Interventions: Drug: lidocaine-Prilocaine cream
- placebo cream (Placebo Comparator): an inert placebo cream placed into their cervix
  Interventions: Drug: placebo cream

INTERVENTIONS:
Drug: lidocaine-Prilocaine cream
  Arms: lidocaine-Prilocaine cream
Drug: placebo cream
  Arms: placebo cream

SUMMARY:
The purpose of the investigators' study was to evaluate whether cervical lidocaine-Prilocaine cream will improve pain scores compared to placebo. The investigators hypothesized that lidocaine-Prilocaine cream will reduce the insertion pain.

DETAILED DESCRIPTION:
IUD can cause pain and discomfort in several ways: Use of the tenaculum to grasp the cervix and straighten the uterus for proper insertion; trans-cervical actions including measuring uterine depth, inserting the IUD insertion tube, and removing the tube; and placement of the device in the uterus.

To minimize the discomfort and the hazards of an IUD insertion, several measures have been proposed including NSAIDs, anxiolytics, and local anesthetics in the form of intracervical gel, cervical and para-cervical block, but there have not done enough studies about their effectiveness. According to the review published in the Cochrane, non-steroidal anti-inflammatory drugs and misoprostol are not effective on reducing an IUD insertion pain. Many trials have been done about effectiveness of lidocaine gel in reducing pain during IUD insertion and only one of those trials showed positive effect of 2% lidocaine gel, while others failed.

Lidocaine 2.5% and Prilocaine 2.5% Cream, is an emulsion in which the oil phase is a eutectic mixture of Lidocaine and Prilocaine cream in a ratio of 1:1 by weight. This eutectic mixture has a melting point below room temperature and therefore both local anesthetics exist as liquid oil rather than as crystals. Its absorption of from the genital mucosa is more rapid and onset time is shorter (5 to 10 minutes) than after application to intact skin. After a 5 to 10 minute application of Lidocaine-Prilocaine cream to female genital mucosa, the average duration of effective analgesia was 15 to 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Women not taken analgesics or anxiolytics in the 24 hours prior insertion
* Women not taken misoprostol prior to IUD insertion
* No contraindication to or history of allergic reaction to lidocaine
* Women who will accept to participate in the study

Exclusion Criteria:

* Lidocaine allergy
* Any contraindication to IUD placement

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Mean pain score during IUD insertion | 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt